CLINICAL TRIAL: NCT01817855
Title: A Phase I, Randomized, DoubleBlind Placebo-Controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Inhaled Doses (MAD) of AZD7624 to Healthy Subjects and Patients With COPD
Brief Title: To Assess the Safety, Tolerability, and Pharmacokinetics of AZD7624 in Healthy Volunteers and COPD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D2550C00002
Record Dates: First submitted 2013-03-18; First posted 2013-03-26 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-02

CONDITIONS: COPD; Healthy Subjects
Keywords: Phase 1,; Safety,; Tolerability,; Healthy,; COPD patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — AZD7624

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Groups 1-4 multiple ascending doses of AZD7624 Healthy subjects will participate in groups 1-3. In each group 6 subjects will receive AZD7624 and 2 will receive matching placebo.
  COPD patients will participate in group 4. In this group, 8 patients will receive AZD7624 and 2 patients will receive matching placebo.
  Interventions: Drug: AZD7624
- 2 (Placebo Comparator): Groups 1-4 multiple ascending doses of placebo Healthy subjects will participate in groups 1-3. In each group 6 subjects will receive AZD7624 and 2 will receive matching placebo.
  COPD patients will participate in group 4. In this group, 8 patients will receive AZD7624 and 2 will receive matching placebo.
  Interventions: Drug: Placebo to match

INTERVENTIONS:
Drug: AZD7624 — Multiple ascending doses (starting from 300 µg lung deposited dose up to 1200 µg) inhaled IMP via a nebulizer
  Arms: 1
Drug: Placebo to match — Multiple doses inhaled placebo via a nebulizer
  Arms: 2

SUMMARY:
This study will investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of AZD7624 in healthy subjects and patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
A Phase I, Randomized, DoubleBlind Placebo-Controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Inhaled Doses (MAD) of AZD7624 to Healthy Subjects and Patients with COPD

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
* Provision of signed and dated, written informed consent prior to any study specific procedures
* Plasma myoglobin and CK not above the upper reference range of the analysing laboratory at Day -1
* Male and/or female patients with COPD aged above18 years with suitable veins for cannulation or repeated venipuncture.
* Clinical diagnosis of COPD for more than 1 year at Visit 1, according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines

Exclusion Criteria:

* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the IP
* Receipt of another new chemical entity (defined as a compound which has not been approved for marketing) or participation in any other clinical study that included drug treatment within at least 3 months of the first administration of the IP in this study
* Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results as judged by the Investigator
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV)
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Khan, MBBS, MRCP, Principal Investigator — Quintiles Drg Research Centre At Guys Hosipital, 6 Newcomen Street London SE1 1YR; Naimish Patel, MD, Study Chair — AstraZeneca, Wilmington, US
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1273&filename=D2550C00002_synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Both the lung deposited doses and total delivered doses are reported in clinical study report, and the conversion is: In cohort 1 to 6, the lung deposited doses 151 µg, 303 µg, 595 µg, 1191 µg, 1160 µg and 580 µg are equivalent to the delivered doses 261µg, 522µg, 1027µg, 2053µg, 1932µg and 966µg, respectively.
Pre-assignment Details: The screening period for all the subjects was from Day -42 to Day -2. Admission on day -1. A 8 to 9 days treatment period, 7 to 9 days follow up period. It was planned to enrol to 32 healthy volunteers and 20 COPD to the study, but 4 COPD patients (Due to stopping cohort 4 prematurly) and one healthy volunteer (in cohort 3) were not enrolled.
Groups:
- AZD7624 Healthy Volunteers: Healthy Volunteers with 261 µg to 2053 µg delivered dose of AZD7624, once daily or twice daily
- Placebo Healthy Volunteers: Healthy Volunteers with Placebo, once daily or twice daily
- AZD7624 COPD: COPD patients with 966 µg or 1932 µg delivered dose of AZD7624, once daily
- Placebo COPD: COPD Patients with Placebo, once daily
Period: Overall Study
Arm/Group | AZD7624 Healthy Volunteers | Placebo Healthy Volunteers | AZD7624 COPD | Placebo COPD
Started | 23 | 8 | 11 | 5
Completed | 23 | 6 | 9 | 5
Not Completed | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least 1 dose of the investigational product, AZD7624 or placebo and for whom any postdose data were available were included in the analysis (safety population).
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD7624 Healthy Volunteers | Placebo Healthy Volunteers | AZD7624 COPD | Placebo COPD | Total
Number analyzed (Participants) | 23 | 8 | 11 | 5 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36 (9.7) | 32 (9.1) | 65 (9.7) | 65 (8.7) | 45.3 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 2 | 3
  Male | 23 | 8 | 10 | 3 | 44

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Summary of number of subjects who had at least one adverse event in any category (Safety analysis set)
Time Frame: Up to 24 days
Measure: Number; unit: Participants
Arm/Group | AZD7624 Healthy Volunteers | Placebo Healthy Volunteers | AZD7624 COPD | Placebo COPD
Number analyzed (Participants) | 23 | 8 | 11 | 5
Participants
  Any Adverse Event (AE) | 6 | 3 | 7 | 2
  Any AE with outcome = death | 0 | 0 | 0 | 0
  Any SAE (including events with outcome = death) | 0 | 0 | 0 | 0
  Any AE leading to discontinuation | 0 | 1 | 2 | 0

2. Secondary Outcome: Summary of Pharmacokinetic Parameters (AUC(0-tau) )
Description: Summary of pharmacokinetic parameters of AZD7624 after multiple once daily dose administration in cohorts 4,5,6 and multiple twice daily administration in cohorts 1,2 and 3, on Days 7, 8 or 9.
  *AUC(0-tau) = AUC(0-last) where for cohorts 2,3,4,5 and 6 tau=24 hours and for cohort 1, tau=12 hours .
  Results are presented for cohort 1,2,3,4,5 with SPIRA device and for cohort 6 with ADI device (test device).
  Number of Participants Analyzed is based on the available data for the used device and for the day that PK measurements were taken.
Time Frame: PK concentration was measured at 0, 15min, 30min, 45min, 1hr, 2hr, 4hr, 6hr, 9hr, 12hr, 18hr and 24hr post dose on Day 7 for cohort 6, Day 8 for cohorts 1,4 and 5 and on Day 9 for cohorts 2 and 3.
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- AZD7624 COPD Cohort 4: COPD patients on Cohort 4 with 1932 µg delivered dose of AZD7624 , once daily
- AZD7624 Healthy Volunteers Cohort 5: Healthy volunteers on Cohort 5 with 2053 µg delivered dose of AZD7624 , once daily
- AZD7624 COPD Cohort 6: COPD patients on Cohort 6 with 966 µg delivered dose of AZD7624, once daily
- AZD7624 Healthy Volunteers Cohort 1: Healthy volunteers on Cohort 1 with 261 µg delivered dose of AZD7624, twice daily
- AZD7624 Healthy Volunteers Cohort 2: Healthy volunteers on Cohort 2 with 522 µg delivered dose of AZD7624, twice daily
- AZD7624 Healthy Volunteers Cohort 3: Healthy volunteers on Cohort 3 with 1027 µg delivered dose of AZD7624, twice daily
Arm/Group | AZD7624 COPD Cohort 4 | AZD7624 Healthy Volunteers Cohort 5 | AZD7624 COPD Cohort 6 | AZD7624 Healthy Volunteers Cohort 1 | AZD7624 Healthy Volunteers Cohort 2 | AZD7624 Healthy Volunteers Cohort 3
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 5
nmol*h/L | 40.1 (11.4) | 27.4 (17.3) | 13.3 (50.4) | 3.88 (28.5) | 9.31 (12.7) | 15.2 (33.3)

3. Secondary Outcome: Summary of Pharmacokinetic Parameters (Cmax)
Description: Summary of pharmacokinetic parameters of AZD7624 after multiple once daily dose administration in cohorts 4,5,6 and multiple twice daily administration in cohorts 1,2 and 3, on Days 7, 8 or 9. Results are presented for cohort 1,2,3,4,5 with SPIRA device and for cohort 6 with ADI device (test device).
  Number of Participants Analyzed is based on the available data for the used device and for the day that PK measurements were taken.
Time Frame: as for outcome 2
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD7624 COPD Cohort 4 | AZD7624 Healthy Volunteers Cohort 5 | AZD7624 COPD Cohort 6 | AZD7624 Healthy Volunteers Cohort 1 | AZD7624 Healthy Volunteers Cohort 2 | AZD7624 Healthy Volunteers Cohort 3
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 5
nmol/L | 11.9 (13.4) | 15.6 (38.3) | 3.08 (54.6) | 2.14 (49.5) | 6.23 (22.8) | 8.07 (39.5)

4. Secondary Outcome: Summary of Pharmacokinetic Parameters (Cmin)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD7624 COPD Cohort 4 | AZD7624 Healthy Volunteers Cohort 5 | AZD7624 COPD Cohort 6 | AZD7624 Healthy Volunteers Cohort 1 | AZD7624 Healthy Volunteers Cohort 2 | AZD7624 Healthy Volunteers Cohort 3
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 5
nmol/L | 0.797 (22.2) | 0.602 (15.7) | 0.355 (47.3) | 0.183 (44.0) | 0.453 (18.6) | 0.719 (36.9)

ADVERSE EVENTS:
Time Frame: Up to 24 days
Arm/Group | AZD7624 Healthy Volunteers | Placebo Healthy Volunteers | AZD7624 COPD | Placebo COPD
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/8 | 0/11 | 0/5
Other Adverse Events (participants affected / at risk) | 6/23 | 3/8 | 7/11 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD7624 Healthy Volunteers (N=23) | Placebo Healthy Volunteers (N=8) | AZD7624 COPD (N=11) | Placebo COPD (N=5)
Cough, Bronchospasm, Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 0
Mouth ulceration, Dry mouth, Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Chest discomfort, Vessel puncture site bruise (General disorders) | 1 | 2 | 2 | 0
Nasopharyngitis, Upper respiratory tract infection, Rhinitis, Tooth abscess (Infections and infestations) | 2 | 1 | 3 | 0
Back Pain, Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Dizziness, Headache, Presyncope (Nervous system disorders) | 0 | 2 | 1 | 1
Papule, Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days